CLINICAL TRIAL: NCT03891368
Title: Randomized Controlled Trial of a Learning Collaborative to Implement Health Promotion in Mental Health
Brief Title: Study of a Learning Collaborative to Implement Health Promotion in Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Dartmouth-Hitchcock Medical Center (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Stephen Bartels, Director, The Mongan Institute, James J. and Jean H. Mongan Chair in Health Policy and Community Health at MGH-Harvard, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH102325 (NIH); R01MH102325 (NIH); STUDY00028067 (Other: Dartmouth College)
Record Dates: First submitted 2019-03-16; First posted 2019-03-27 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-08

CONDITIONS: Health Promotion; Obesity; Organizational Innovation; Mental Health Services
Keywords: Learning collaborative; Technical assistance; Serious mental illness; Organizational change; InSHAPE
MeSH Terms: conditions — Obesity | interventions — Health Planning Technical Assistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Learning Collaborative (Experimental): The virtual learning collaborative (VLC) is an 18-month intensive training, skill building, and structured implementation process focused on reinforcing fidelity to the InSHAPE model.
  Interventions: Other: Virtual Learning Collaborative
- Technical Assistance (Active Comparator): The technical assistance (TA) condition includes four scheduled conference calls between an InSHAPE expert TA "coach" and the agency's InSHAPE team, with the option for sites to request additional calls as needed through 18-months post-randomization.
  Interventions: Other: Technical Assistance

INTERVENTIONS:
Other: Virtual Learning Collaborative — InSHAPE teams consisting of health mentors, supervisors, and senior leaders from each mental health agency randomized to the VLC will be invited to attend an in-person initial kick-off meeting followed by once per month 90-minute VLC sessions. The VLC is organized into three stages: Prework, Action, and Continuous Improvement. VLC faculty, including interventionists with expertise in implementation science, quality improvement, and subject matter (i.e., InSHAPE) experts, will facilitate VLC sessions following a structured protocol to standardize the planning and execution of the VLC across three cohorts enrolled in the study.
  Arms: Virtual Learning Collaborative
Other: Technical Assistance — Scheduled calls will occur at 1 month, 2 months, 8 months, and 14 months following their participation in initial InSHAPE training following randomization and follow a structured protocol. At the end of each scheduled conference call, the coach will schedule the next call with the site.
  Arms: Technical Assistance

SUMMARY:
Healthcare organizations have increasingly formed quality-improvement Learning Collaboratives to improve care for specific populations; however, there are few data on the effectiveness of this strategy compared to conventional training approaches. The primary aim of this cluster randomized implementation trial is to evaluate the effectiveness of a virtual learning collaborative (VLC) in the implementation of a lifestyle intervention for persons with serious mental illness (SMI) in routine mental health settings, compared to typical implementation consisting of site training and one-on-one individual technical assistance (TA). The investigators hypothesize that VLC compared to TA will be associated with greater Program Participation, Program Fidelity, and a greater proportion of participants achieving clinically significant weight loss.

DETAILED DESCRIPTION:
Despite the existence of a variety of evidence-based health promotion practices, it is not well documented how to effectively transform community mental health organizations to embrace wellness as central to their mission and services. Healthcare organizations have increasingly formed quality-improvement Learning Collaboratives to improve care for specific populations; however, there are few data on the effectiveness of this strategy compared to conventional training approaches. The primary aim of this cluster randomized implementation trial is to evaluate the effectiveness of a virtual learning collaborative (VLC) in the implementation of a lifestyle intervention for persons with serious mental illness (SMI) in routine mental health settings, compared to typical implementation consisting of site training and one-on-one individual technical assistance (TA). Forty-eight mental health provider organizations from across the United States providing behavioral health services to people with SMI will be recruited to participate in collaboration with the National Council for Behavioral Health. The evidence-based practice to be implemented is the InSHAPE health coaching intervention for persons with SMI. Sites will be stratified by size and randomized to receive an 18-month intensive group-based VLC with monthly learning sessions or individual technical assistance with four scheduled conference calls over 18 months. Sites will be enrolled in three blocks of 16 sites each. The investigators will compare implementation VLC to TA with respect to service outcomes, implementation outcomes, and participant outcomes:

Aim 1 (Service Outcomes): Compare the effectiveness of VLC to TA with respect to Program Participation as measured by the proportion of enrolled individuals who received an adequate exposure to the evidence-based practice, as defined by attending at least 50% of the InSHAPE Health Mentor sessions over 6 months.

(H1) Hypothesis: VLC compared to TA will be associated with greater Program Participation.

Aim 2 (Implementation Outcomes): Compare VLC to TA with respect to Program Fidelity as measured by the InSHAPE Fidelity Scale.

(H2) Hypothesis: VLC compared to TA will be associated with greater Program Fidelity.

Aim 3 (Participant Outcomes): Compare VLC to TA with respect to adult participants with SMI enrolled in the InSHAPE program achieving clinically significant weight loss (≥5% weight loss).

(H3) Hypothesis: VLC compared to TA will be associated with a greater proportion of InSHAPE participants achieving clinically significant weight loss.

Secondary aims:

The investigators will also examine the following exploratory hypotheses: VLC compared to TA will result in (E1) more rapid Full Program Operation; (E2) greater Program Uptake; (E3) significantly improved participant health behaviors of physical activity and nutrition; and (E4) greater likelihood of Program Sustainability at 24 months. The investigators will also explore (E5) the effect of Organizational Change and VLC fidelity on Program Participation, and (E6) agency participation and adherence to the core elements of a Learning Collaborative as a predictor of InSHAPE program participation, InSHAPE program fidelity, and participant weight outcomes.

ELIGIBILITY:
Mental Health Provider Organizations Inclusion Criteria:

* Provide outpatient behavioral health services to people with SMI as defined by primary DSM-V Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder or any other state-certified serious mental illness diagnosis (e.g., post-traumatic stress disorder)
* Agree to study procedures including a commitment by CEO or designee to: (a) participate over the full program, including randomization to VLC or TA; (b) engage (if randomized to VLC) in monthly web-based meetings with other VLC members, including sharing implementation outcome data and performance evaluations; (c) collect and submit aggregate participant-level data, including demographics, weight/BMI, physical fitness as measured by a 6-minute walk test, waist circumference, frequency of physical activity, and self-reported changes in nutrition; and (d) participate in phone-based organizational change and implementation assessments, including organization leadership, middle management, and InSHAPE staff.

InSHAPE Participant Inclusion Criteria:

* Age 18 or older
* SMI as defined by primary DSM-V Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder or any other state-certified SMI diagnosis (e.g., post-traumatic stress disorder)
* Verbal permission from participant to share de-identified data with the research team
* Overweight or obesity as indicated by BMI of 25 kg/m2 or greater
* Medical clearance for participation in an exercise and dietary medication program by a physician, physician assistant, or nurse practitioner.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Program Participation | 6, 12, 18, and 24 months
  Program Participation will be measured as the proportion of InHAPE participants who have been enrolled and have received adequate exposure to the intervention, defined by attending at least 50% of health mentor sessions over 6 months.
Change in Program Fidelity | 6, 12, and 24 months
  Program Fidelity will be measured using the 22-item InSHAPE Fidelity Scale which assesses structural elements of program implementation in the domains of staffing, organization, and services. Items are rated on a 5-point behaviorally-anchored scale ranging from 1 (not implemented) to 5 (fully implemented) (e.g., weekly review of exercise objectives is scored 5 if 90-100% of required exercise logs are completed, a score of 1 represents 0-24%). The 22 items give a total score ranging from 22 to 110, with a higher score indicating stronger fidelity to the InSHAPE model.
Change in Participant Weight | Baseline, quarterly through 24 months
  Participant Weight will be defined as clinically significant weight loss of ≥5% body weight since baseline, and weight will be measured to the tenth of a pound on a digital bathroom scale.

SECONDARY OUTCOMES:
Change in Full Program Operation defined as a 1.0 FTE Health Mentor with a caseload of 20 participants | 12 and 24 months
  Full Program Operation will be measured by time to having 1.0 FTE Health Mentor with a caseload of 20 participants.
Change in Program Uptake defined as the number of 1.0 FTE Health Mentors | 12 and 24 months
  Program Uptake will be measured by the number of 1.0 FTE Health Mentors and participants served at 12 and 24 months.
Change in Participant Cardiorespiratory Fitness | Baseline, quarterly through 24 months
  Participant Cardiorespiratory Fitness will be assessed using the 6-Minute Walk Test, which measures the distance an individual can walk in six minutes. An increase in distance of >50 meters on the 6-MWT is associated with clinically significant reduction in risk for cardiovascular disease.
Change in Participant Dietary Behavior | Baseline, quarterly through 24 months
  Participant Dietary Behavior will be assessed using Weight Loss Behavior Stages of Change Scale. Higher scores indicate greater readiness to change dietary behaviors. An overall dietary behavior score consisting of the mean for the items related to three domains: portion control, consumption of dietary fat, and intake of fruits and vegetables will be calculated.
Change in Participant Physical Activity | Baseline, quarterly through 24 months
  Participant Physical Activity will be assessed using the short-form International Physical Activity Questionnaire. Summary scores will be calculated for vigorous activities obtaining an estimate of weekly metabolic equivalent expenditure (MET) minutes of vigorous physical activity.
Change in Program Sustainability defined as having a Health Mentor who meets with at least one InSHAPE participant | 24 months
  Program Sustainability at 24-month follow-up will be measured by the number of sites still implementing InSHAPE, as defined by having a Health Mentor who has a personal trainer certification and who meets with at least one InSHAPE participant.
Change in Organizational Change that supports an organization's capacity to implement and sustain the InSHAPE program | 3, 12, and 24 months
  Organizational Change will be measured using the Dartmouth Organizational Structure Scale (DOSS), an 11-item interviewer-rated scale developed by the investigators. It measures a set of practices and procedures aimed at supporting the organization's capacity to implement and sustain the InSHAPE program. The content dimensions include leadership, financing, policies, agency commitment to the evidence-based practice, process and outcome monitoring for quality improvement, and other organizational factors found in prior implementation studies to be associated with successful implementation of evidence-based practices. Each DOSS item is scored on a 5-point behavioral-anchored continuum. The interviewer assesses five objective criteria for each item, giving one point for each criterion met for a maximum score of 5. The 11 items are summed, yielding a total DOSS score with possible values ranging from 11 to 55, with a higher score indicating greater organizational change.
Change in VLC Adherence | Up to 18 months
  VLC Adherence will be measured using an 11-item VLC Adherence Tool. The tool was developed by the investigators for the study based on a review of the literature, feedback from experts and the research team, and feasibility testing. Key domains include the extent to which a team engages in verbal participation, chat box participation, implementation progress, use of quality improvement tools or approaches, use of data collection to drive improvement, collaborative learning and sharing, and planning for program sustainment. VLC faculty score each team on every domain by consensus at the conclusion of each learning session based on a review of submitted homework, participation, and group interaction. Total score ranges from 0 (poor VLC adherence) to 41 (strong VLC adherence).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bartels, MD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Derived] Aschbrenner KA, Pratt SI, Bond GR, Zubkoff L, Naslund JA, Jue K, Williams G, Kinney A, Cohen MJ, Godfrey MM, Bartels SJ. A virtual learning collaborative to implement health promotion in routine mental health settings: Protocol for a cluster randomized trial. Contemp Clin Trials. 2019 Sep;84:105816. doi: 10.1016/j.cct.2019.105816. Epub 2019 Jul 22. PMID 31344520